CLINICAL TRIAL: NCT06455332
Title: Evaluation of the Predictive Value of the Optic Nerve Involvement at the Stage of Clinically Isolated Syndrome, for the Diagnosis of Clinically Definite Multiple Sclerosis and the Delay of Second Relapses' Occurrence
Brief Title: Predictive Value of the Optic Nerve Involvement in Clinically Isolated Syndrome
Acronym: HdeFIMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Région Nord-Pas de Calais, France (Other); Amiens University Hospital (Other); Boulogne sur Mer Hospital Center (Other); Centre Hospitalier VALENCIENNES (Other); Centre Hospitalier de Roubaix (Other); Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021_0474
Record Dates: First submitted 2024-05-23; First posted 2024-06-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Clinically Isolated Syndrome; Multiple Sclerosis
Keywords: Clinically isolated syndrome; Multiple sclerosis; MRI; Optical coherence tomography; Optic nerve; Diagnostic criteria
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients will part of the same follow-up study. (Experimental): All patients will part of the same follow-up study. No treatment will be compared. Patients will be treated as recommended.
  Interventions: Other: Optic nerve MRI sequence

INTERVENTIONS:
Other: Optic nerve MRI sequence — Systematic optic nerve MRI sequence during the CIS diagnosis work-up. This sequence is not done systematically and not recommended for now (except in case of acute ON). The interventional nature of the study remains minimal

SUMMARY:
Optic neuritis (ON) represents around 30% of clinical presentation of clinically isolated syndrome (CIS). Asymptomatic optic nerve involvement is very frequent in all stage of multiple sclerosis (MS) disease including the CIS. However, optic nerve is still not part of MS diagnosis criteria. The main objective of our regional and multicenter study is to evaluate the prognostic value of optic nerve involvement at the earliest clinical stage of MS (=CIS) for the diagnosis of clinically definite MS (2nd clinical relapse) and the delay until the 2nd relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 55 years old
* Occurrence of CIS ≤ 6 months
* With two T2 hypersignals on brain/spinal cord MRI suggestive of MS or with oligoclonal bands
* Giving their written informed consent

Exclusion Criteria:

* Pathological conditions that may skew the optic nerve MRI and/or retinal OCT (diabetes mellitus, glaucoma, retinopathy, ametropia >6 dioptria)
* Past history of MS relapses
* Extensive myelitis (>3 vertebral bodies)
* Bilateral optic neuritis without T2 lesions suggestive of MS
* Contra-indication to MRI, gadolinium injection
* Pregnancy, breast-feeding
* Patients unable to consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Optic nerve involvement defined by occurrence of a recent clinical episode of ON | assessed at baseline
Asymptomatic optic nerve involvement defined by MRI (detection of an optic nerve T2 hypersignal) | assessed at baseline
Risk of a new clinical relapse will be assessed by the occurrence and time to onset of a second MS clinical relapse | assessed every 6 months during 24 months
Asymptomatic optic nerve involvement defined by OCT (GCIPL-IETD,3pm) | assessed at baseline
Risk of a new clinical relapse will be assessed by the occurrence and time to onset of a CDMS | assessed every 6 months during 24 months

SECONDARY OUTCOMES:
Asymptomatic optic nerve involvement will be defined by: - asymptomatic optic nerve T2 hypersignal detected on one or both optic nerve(s) - or by GCIPL-IETD,3pm measured by OCT - or by GCIPL-IETD≥3µm measured by OCT | assessed at baseline every 6 months during 24 months
  Time to the second clinical relapse occurrence will be assessed every 6 months during 24 months at each neurological examination (M0, M6, M12, M18, M24)
Time to the second clinical relapse occurrence will be assessed every 6 months during 24 months at each neurological examination | assessed at Month 0, Month 6, Month 12, Month 18, Month 24

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Roger Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No